CLINICAL TRIAL: NCT07069179
Title: Choose to Move Replacement Ready: A Feasibility Trial of a Virtual Health-promoting Intervention for People Awaiting Total Hip or Knee Replacement Surgery
Brief Title: Feasibility of Choose to Move Replacement Ready
Acronym: CTM-RR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Active Aging Society (Other); Specialist Services Committee (Doctors of BC) (Unknown)
Responsible Party: Principal Investigator, Heather McKay, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H24-03805
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis; Osteoarthritis (OA) of the Knee; Osteoarthritis, Hip; Total Knee Arthroplasty; Total Hip Arthroplasty; Mobility Limitation; Social Isolation or Loneliness; Pain; Implementation Science; Physical Inactivity; Sedentary Behaviors
Keywords: Osteoarthritis; Implementation science; Social isolation; Physical activity; Mobility; Loneliness; Pain; Joint replacement; Feasibility; Acceptability; Fidelity
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip; Mobility Limitation; Social Isolation; Pain; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Choose to Move Replacement Ready (Experimental): CTM-RR is a 3-month program for individuals with hip and/or knee osteoarthritis on surgical waitlists for total hip or total knee replacement that includes three required components: 1) a 30-min one-on-one virtual consultation (via Zoom) where activity coaches support participants to set goals and develop a PA action plan; 2) 8 virtual group meetings (via Zoom, 90-min each) facilitated by activity coaches, with small groups of participants (10/program) who provide peer support. Each meeting includes: i) two, 15-min movement breaks where participants perform structured hip and knee exercises delivered by the coach and ii) education and discussion on relevant topics (e.g. goal setting, PA, what to expect from surgery); 3) Home-based hip and knee exercises to complete independently, 2x/week. Optional components of CTM-RR include 4) a bi-weekly newsletter distributed by the AAS and 5) peer support check-ins outside of group meetings.
  Interventions: Behavioral: Choose to Move Replacement Ready

INTERVENTIONS:
Behavioral: Choose to Move Replacement Ready — As described under study arm description.

SUMMARY:
Choose to Move (CTM) is a 3-month, choice-based health-promoting program for low active older adults being scaled-up across British Columbia (BC), Canada. Recently, the investigators adapted CTM for the >14000 people in BC who are on surgical waitlists for total knee replacement or total hip replacement (TKR/THR) for osteoarthritis (OA). The primary goal of this observational study is to learn if the adapted program, Choose to Move Replacement Ready (CTM-RR), is feasible to deliver to people with hip and/or knee osteoarthritis who are on surgical waitlists for TKR/THR.

Participants who enrol in CTM-RR will answer online survey questions about the program and about their physical activity, mobility, pain, function, quality of life, willingness to undergo surgery, overall perception of their joint condition, psychosocial health, self-efficacy, social isolation, loneliness, and sedentary time. CTM-RR activity coaches will also answer online survey questions about the program. CTM-RR participants, activity coaches, and referral partners will also participate in interviews about the program.

DETAILED DESCRIPTION:
Choose to Move (CTM) an effective 3-month, choice-based health-promoting program for low active older adults being scaled-up in phases across British Columbia (BC), Canada. Choose to Move Replacement Ready (CTM-RR) is an adapted version of the program tailored to support individuals with hip and/or knee osteoarthritis on surgical waitlists for TKR/THR, with the overall goal of enhancing key health outcomes. Trained activity coaches hired by the Active Aging Society will deliver CTM-RR to individuals on surgical waitlists for TKR/THR. The investigators will then evaluate implementation of CTM-RR, and the impact of CTM-RR on participants' physical and social health.

The primary objective of this trial is to:

1. Assess implementation outcomes (participant recruitment, retention, dose delivered/received, fidelity) of the adapted CTM model against predetermined feasibility targets.

   The secondary objectives are to:
2. Describe implementation determinants (acceptability, feasibility, appropriateness) and outcomes (reach, adaptations, perceived participant responsiveness, adoption) of the adapted CTM model.
3. Evaluate the preliminary estimates of effectiveness of CTM-RR. Specifically, whether CTM-RR increases participants' pre-operative moderate-to-vigorous physical activity, light physical activity, mobility, psychosocial health, and self-efficacy to manage their condition; improves their perception of their joint condition, function, and quality of life; and decreases pain, social isolation, loneliness, and sedentary time
4. Assess whether participant-level health benefits, if any, are maintained 6 months after participants complete the CTM-RR program.

In partnership with the Active Aging Society, the investigators aim to deliver 6 CTM-RR online programs over 9-months to approximately 60 participants total across BC. There is no cost to participate in the CTM-RR program, and individuals may participate in CTM-RR regardless of whether they choose to be evaluated as part of this trial.

The investigators will conduct a feasibility trial using a hybrid implementation-effectiveness type 2 trial design. Data will be collected at 0 (baseline), 3 (post-intervention), and 9 (long-term follow-up) months to assess implementation and impact of CTM-RR, and maintenance of any program-related benefits. The investigators will also collect physical activity logs from program participants (weekly, during program participation).

ELIGIBILITY:
Inclusion Criteria:

1. Activity coach hired by the Active Aging Society (activity coaches must speak English to participate in the evaluation);
2. English-speaking older adults (aged >=50 years) who participate in CTM-RR will be invited to participate in the evaluation
3. Referral partner (People who work in a healthcare setting who refer patients into the program)

Exclusion Criteria:

1. non-English speaking activity coach
2. non-English speaking referral partner

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Implementation Outcome: Recruitment | baseline
  Obtained from program records. Proportion of people who attend the program information session, are eligible, and enrol in the program.
  Feasibility Target: Enrol 50% of people attending the program information session who are eligible to participate to the program.
Implementation Outcome: Retention | baseline, 3, 9 months
  Obtained from evaluation records. Proportion of participants who consent to the evaluation who complete each follow-up assessment.
  Feasibility target: A minimum of 80% of participants who consented to the evaluation (and are in the pre-operative period) completing each follow-up assessment.
Implementation Outcome: Dose delivered | 3 months
  Obtained from post-program survey. Proportion of required intervention components (group meetings and one-on-one consultations) delivered by activity coaches.
  Feasibility target: Activity coaches delivering 90% of required intervention components (group meetings and one-on-one consultations).
Implementation Outcome: Dose received | 3 months
  Obtained from post-program survey. Proportion of participants who consent to the evaluation, attending required intervention components (group meetings and one-on-one consultation)
  Feasibility target: Participants who consent to the evaluation attending 6 out of 9 (>60%) of required intervention components (group meetings and one-on-one consultation)
Implementation Outcome: Fidelity (Proportion of participants who adhered to prescribed exercise) | 3 months
  Obtained from post-program survey. Measures adherence to prescribed frequency, intensity, duration, and type of exercises performed.
  80% of participants adhered to all of the following criteria:
  * on average, frequency= two sessions per week or greater
  * on average, intensity= 7 out of 10 rating of perceived exertion or greater
  * on average, duration= 20 minutes or greater
  * on average, exercises were completed as prescribed without omission or substitution of prescribed exercises
Adverse events: Number of adverse events | 3 months
  Obtained from post-program survey. Number of adverse events related to Choose to Move: Replacement Ready that required medical treatment and/or lasted two or more days.

SECONDARY OUTCOMES:
Change in physical activity | baseline, 3, 9 months
  Single-item physical activity questionnaire. Output measure is self-reported number of days engaging in ≥30 minutes of moderate-to-vigorous physical activity in the past week (range 0-7). Higher scores reflect a better outcome (i.e. increased physical activity)
Change in light physical activity | baseline, 3, 9 months
  International Physical Activity Questionnaire (IPAQ-SF): assesses self-reported weekly minutes of light physical activity (MET minutes per week)
Change in sedentary time | baseline, 3, 9 months
  International Physical Activity Questionnaire (IPAQ-SF): assesses self-reported weekly minutes of sedentary time
Change in bone and muscle strengthening activity | baseline, 3, 9 months
  Single-item muscle strengthening activity survey. Number of days in past week doing activities that increase bone and muscle strength
Change in balance activity | baseline, 3, 9 months
  Single-item activity survey. Number of days in past week doing activities that improve balance.
Change in capacity for mobility | baseline, 3, 9 months
  Short-Form-36 health survey (SF-36) Physical Functioning Scale: two items assess self-reported ability to walk ¼ mile and 1 flight of stairs.
Change in social isolation | baseline, 3, 9 months
  Social Isolation Questionnaire: score (0-15) reflects the degree of social interaction and support. Higher scores indicate a greater level of social interaction and support.
Change in loneliness | baseline, 3, 9 months
  The 3-item U.S. Health and Retirement Study Participant Lifestyle Questionnaire reflects experiences of loneliness. Each item is scored on a scale of 1-3. The output variable is the summed score of the 3 items (range 3-9); Higher scores indicate greater perceived loneliness.
Change in ability to participate in daily activities | baseline, 3, 9 months
  The four-item PROMIS- Ability to Participate in Social Roles and Activities Scale- short form 4a will be used to assess perceived ability to perform one's usual social roles and activities. Each item is scored on a scale of 1-5. The output variable is the summed raw score of all 4-items (range 4-20) converted into a T-score (27.5-64.2) ; higher scores indicate greater ability to engage in social roles and activities.
Change in Hip disability and Osteoarthritis Outcome 12-item Score | baseline, 3, 9 months
  The 12-item Hip Disability and Osteoarthritis Outcome Score (HOOS-12) assesses patients' hip condition (pain, function, quality of life). Each item is scored on a scale of 0-10. The output variable is the average score of the 12-items (range 0-100); higher scores indicate worse hip problems.
Change in Knee disability and Osteoarthritis Outcome 12-item Score | baseline, 3, 9 months
  The 12-item Knee Disability and Osteoarthritis Outcome Score (KOOS-12) assesses patients' knee condition (pain, function, quality of life). Each item is scored on a scale of 0-10. The output variable is the average score of the 12-items (range 0-100); higher scores indicate worse knee problems.
Change in patient global assessment of target joint | baseline, 3, 9 months
  Single-item measure using a numerical rating scale: score (0-10) assesses the overall condition of the affected hip or knee joint. Higher scores indicate worse condition (severe symptoms).
Change in arthritis-specific self-efficacy | baseline, 3, 9 months
  The 8-item questionnaire assesses how certain an individual is that they can manage various aspects of their arthritis. Each item is scored on a scale of 1-10. The output variable is the average score of all 8-items (range 8-80); higher scores indicate more self-efficacy.
Change in pain intensity | baseline, 3, 9 months
  Pain Numerical Rating Scale (NRS): score (0-10) assesses pain intensity on average during the past week. Higher scores indicate worse pain intensity.
Change in willingness to undergo surgery | baseline, 3, 9 months
  One item will assess participants' willingness to undergo hip or knee replacement surgery. The question asks: "What is your current willingness to undergo a [total hip replacement surgery or total knee replacement surgery]?" The response options are: definitely unwilling, probably unwilling, unsure, probably willing or definitely willing. Definitely unwilling, probably unwilling, unsure= No, and probably willing or definitely willing=Yes. The output variable is self-reported willingness to undergo surgery (yes/no).
Change in anxiety | baseline, 3, 9 months
  The Generalized Anxiety Disorder 7-item scale (GAD-7) will be used to assess the presence of anxiety. Each item is scored on a scale of 0-3. The output variable is the summed total of all scores (range 0-21); higher scores indicate greater levels of anxiety.
Change in kinesiophobia | baseline, 3, 9 months
  The 11-item Tampa Scale for Kinesiophobia (TSK-11) assesses fear of movement in individuals with chronic pain. Each item is scored on a scale of 1-4. The output variable is the total summed score of all 11-items (range 11-44); higher scores indicate greater fear of movement.

OTHER OUTCOMES:
Acceptability - CTM-RR program | 3 months
  Acceptability of Intervention Measure (AIM). Activity coaches' perception that CTM-RR is agreeable or satisfactory will be assessed by survey (4 items each on a 1-5 Likert scale with 1 being completely disagree and 5 being completely agree).
Appropriateness - CTM-RR program | 3 months
  Intervention Appropriateness Measure (IAM). Extent to which CTM-RR fits the needs of the target population will be assessed by survey (4 items each on a 1-5 Likert scale with 1 being completely disagree and 5 being completely agree)
Feasibility - CTM-RR program | 3 months
  Feasibility of Intervention Measure (FIM). Activity coaches' perception that CTM-RR is feasible to deliver will be assessed by survey (4 items each on a 1-5 Likert scale with 1 being completely disagree and 5 being completely agree).
Reach | 3 months
  Number of individuals participating in CTM-RR programs will be obtained from program records.
Adoption | baseline
  Obtained from program records. Number of referral partners who refer participants to the program.
Satisfaction with CTM-RR (survey) | 3 months
  Satisfaction with CTM-RR will be assessed via participant (older adults) survey (designed in house). Higher scores (1-5 Likert scale) indicate higher participant satisfaction with the intervention.
Perceived participant responsiveness (survey) | 3 months
  Perceived participant responsiveness will be assessed via participant (older adults) survey ( short answer responses; developed in house). Older adults will indicate which optional intervention components they engaged in (peer check-in, e-mail newsletter, hip and knee exercises; yes/no response options)
Adaptation (survey) | 3 months
  Planned or purposeful changes to the delivery of CTM-RR by activity coaches will be assessed by survey (short answer responses; developed in house). Coaches will indicate if they made any adaptations to the program (yes/no) and to provide details of any adaptations such as why it needed to occur.
Perceived participant responsiveness (survey) | 3 months
  Perceived participant responsiveness will be assessed via participant (activity coach) survey (developed in house). Activity coaches will indicate whether participants were interactive, enthusiastic, interested, and engaged during group meetings.
Adaptation (interview) | 3 months
  Planned or purposeful changes to the delivery of CTM-RR by activity coaches will be assessed by interview.
Experience with training and program delivery (interview) | 3 months
  Activity coaches overall experience with program training and delivery, will be assessed by interview
Perceived participant responsiveness (interview) | 3 months
  Activity coaches perceptions of participant responsiveness will be assessed by interview.
Adaptations (interview) | 3 months
  Older adults' perceptions of potential adaptations to improve the program will be assessed by interview
Perceived participant responsiveness (interview) | 3 months
  Older adults' responsiveness during the program will be assessed by interview.
Acceptability- CTM-RR program (interview) | 3 months
  Older adults' perceptions that the program is acceptable or satisfactory will be assessed by interview.
Feasibility- CTM-RR program (interview) | 3 months
  Older adults' perceptions of the program's feasibility will be assessed by interview.
Appropriateness- CTM-RR program (interview) | 3 months
  Older adults' perceptions of the program's appropriateness will be assessed by interview.
Feasibility - CTM-RR referral process (interview) | 3 months
  Referral partners' perception that the CTM-RR referral process can be used successfully within the organization will be assessed by interview.
Acceptability - CTM-RR referral process (interview) | 3 months
  Referral partners' perception that the CTM-RR referral process is acceptable or satisfactory will be assessed by interview.
Appropriateness - CTM-RR referral process (interview) | 3 months
  Referral partners' perception regarding the extent to which the CTM-RR referral process fits with the mission, priorities, and values of the organization will be assessed by interview.
Physical activity goal setting | baseline
  At the start of the program, older adult participants complete an Action Plan with support from their activity coach. They record a physical activity goal that is specific, measurable, attainable, relevant, and time-based (SMART). Action Plans will be collected and information from the Action Plans will be reported descriptively.
Self-reported physical activity participation | Weekly (from baseline to 3 months)
  Older adult participants will record the type and duration of physical activities they engaged in over the past 7 days on a weekly basis during CTM-RR. Data will be reported descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A. McKay, PhD, Principal Investigator — University of British Columbia; Laura Churchill, PT, PhD, Principal Investigator — University of British Columbia; Joanie Sims Gould, MSW, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Active Aging Research Team, Robert H. N. Ho Research Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peer MA, Lane J. The Knee Injury and Osteoarthritis Outcome Score (KOOS): a review of its psychometric properties in people undergoing total knee arthroplasty. J Orthop Sports Phys Ther. 2013 Jan;43(1):20-8. doi: 10.2519/jospt.2013.4057. Epub 2012 Dec 7. PMID 23221356
- [Background] Nilsdotter AK, Lohmander LS, Klassbo M, Roos EM. Hip disability and osteoarthritis outcome score (HOOS)--validity and responsiveness in total hip replacement. BMC Musculoskelet Disord. 2003 May 30;4:10. doi: 10.1186/1471-2474-4-10. Epub 2003 May 30. PMID 12777182
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Hawker GA, Bohm E, Dunbar MJ, Faris P, Jones CA, Noseworthy T, Ravi B, Woodhouse LJ, Marshall DA; BEST-Knee Study Team. Patient appropriateness for total knee arthroplasty and predicted probability of a good outcome. RMD Open. 2023 Apr;9(2):e002808. doi: 10.1136/rmdopen-2022-002808. PMID 37068914
- [Background] Alghadir AH, Anwer S, Iqbal A, Iqbal ZA. Test-retest reliability, validity, and minimum detectable change of visual analog, numerical rating, and verbal rating scales for measurement of osteoarthritic knee pain. J Pain Res. 2018 Apr 26;11:851-856. doi: 10.2147/JPR.S158847. eCollection 2018. PMID 29731662
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Klassbo M, Larsson E, Mannevik E. Hip disability and osteoarthritis outcome score. An extension of the Western Ontario and McMaster Universities Osteoarthritis Index. Scand J Rheumatol. 2003;32(1):46-51. doi: 10.1080/03009740310000409. PMID 12635946
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Durlak JA, DuPre EP. Implementation matters: a review of research on the influence of implementation on program outcomes and the factors affecting implementation. Am J Community Psychol. 2008 Jun;41(3-4):327-50. doi: 10.1007/s10464-008-9165-0. PMID 18322790
- [Background] McKay H, Naylor PJ, Lau E, Gray SM, Wolfenden L, Milat A, Bauman A, Race D, Nettlefold L, Sims-Gould J. Implementation and scale-up of physical activity and behavioural nutrition interventions: an evaluation roadmap. Int J Behav Nutr Phys Act. 2019 Nov 7;16(1):102. doi: 10.1186/s12966-019-0868-4. PMID 31699095
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Bauer GR, Braimoh J, Scheim AI, Dharma C. Transgender-inclusive measures of sex/gender for population surveys: Mixed-methods evaluation and recommendations. PLoS One. 2017 May 25;12(5):e0178043. doi: 10.1371/journal.pone.0178043. eCollection 2017. PMID 28542498
- [Background] Veroff JB. The dynamics of help-seeking in men and women: a national survey study. Psychiatry. 1981 Aug;44(3):189-200. PMID 7267859
- [Background] Simonsick EM, Newman AB, Visser M, Goodpaster B, Kritchevsky SB, Rubin S, Nevitt MC, Harris TB; Health, Aging and Body Composition Study. Mobility limitation in self-described well-functioning older adults: importance of endurance walk testing. J Gerontol A Biol Sci Med Sci. 2008 Aug;63(8):841-7. doi: 10.1093/gerona/63.8.841. PMID 18772472
- [Background] Macdonald HM, Nettlefold L, Bauman A, Sims-Gould J, McKay HA. Pragmatic Evaluation of Older Adults' Physical Activity in Scale-Up Studies: Is the Single-Item Measure a Reasonable Option? J Aging Phys Act. 2022 Feb 1;30(1):25-32. doi: 10.1123/japa.2020-0412. Epub 2021 Aug 4. PMID 34348228
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Milton K, Bull FC, Bauman A. Reliability and validity testing of a single-item physical activity measure. Br J Sports Med. 2011 Mar;45(3):203-8. doi: 10.1136/bjsm.2009.068395. Epub 2010 May 19. PMID 20484314
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- See also: Choose to Move website — https://choosetomove.ca
- See also: Active Aging Research Team website — https://activeagingrt.ca
- See also: Aging Aging Society website — https://www.activeagingsociety.org